CLINICAL TRIAL: NCT01387802
Title: Canadian Humira Post Marketing Observational Epidemiological Study: Assessing Effectiveness in Ankylosing Spondylitis (Complete - AS)
Brief Title: Canadian Humira Post Marketing Observational Epidemiological Study: Assessing Effectiveness in Ankylosing Spondylitis
Acronym: Complete-AS
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: JSS Medical Research Inc. (Industry); Cato Research (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-672
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Ankylosing Spondylitis
Keywords: Assessing Effectiveness in Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-Biologic arm: Patients that have not responded to the current treatment with an NSAID (Nonsteroidal Anti-Inflammatory Drug) and/or non - biologic DMARD (Disease-Modifying Anti Rheumatic Drug) for peripheral joint involvement and switch to or addition of another NSAID /DMARDS
- Biologic arm: Patients that have not responded to the current treatment with non biologic DMARDS (Disease-Modifying Anti Rheumatic Drug) /NSAID (Nonsteroidal Anti-Inflammatory Drug) and switch to or addition of adalimumab

SUMMARY:
The current study will assess the real - life effectiveness of adalimumab in the management of Ankylosing Spondylitis (AS) with emphasis on the prevention and management of extra-articular manifestations.

ELIGIBILITY:
Inclusion Criteria:

* Adult >= 18 years old
* Has provided written informed consent allowing the use of their data for the study and providing permission for contact by the study personnel
* Active Ankylosing Spondylitis as per the judgment of the treating physician
* Inadequate response or non tolerant to current NSAID (Nonsteroidal Anti-Inflammatory Drug) or DMARD (Disease-Modifying Anti Rheumatic Drug) based treatment for AS

Exclusion Criteria:

* Currently participating in another prospective study including controlled clinical trials and observational studies
* Patient cannot or will not sign informed consent
* Stable disease with adequate tolerance and response to current treatment and no change in treatment is indicated
* Previous treatment with anti-TNF (Tumor Necrosis Factor) or other biologic agent
* Presence of other condition that, in the opinion of the treating physician, prohibits the patient from participating in the study or obscures the assessment of the treatment of AS

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Offices of community rheumatologists
Sampling Method: Non-Probability Sample
Enrollment: 722 (Actual)
Dates: Start 2011-06-29 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Occurrence, flare-up or exacerbation of Extra Articular Manifestations in Uveitis | Every 3 months up to 6 months, then every 6 months up to 24 months
  Baseline will be assessed as follows: Never Present, Positive History (Not present- Complete Remission,Time since remission onset; Present- Assessment of severity using a five point Likert scale (0 = Absent (Clear for Psoriasis); 5 = Most Severe)) Follow-up visits will be assessed as follows:Not present (Never present, Complete remission) Present (New Onset or Recurrence, Assessment of severity using a five point Likert scale (0 = Absent; 5 = Most Severe))
Occurrence, flare-up or exacerbation of Extra Articular Manifestations in Psoriasis | Every 3 months up to 6 months, then every 6 months up to 24 months
  Baseline will be assessed as follows: Never Present, Positive History (Not present- Complete Remission,Time since remission onset; Present- Assessment of severity using a five point Likert scale (0 = Absent (Clear for Psoriasis); 5 = Most Severe)) Follow-up visits will be assessed as follows:Not present (Never present, Complete remission) Present (New Onset or Recurrence, Assessment of severity using a five point Likert scale (0 = Absent; 5 = Most Severe))
Occurrence, flare-up or exacerbation of Extra Articular Manifestations in Inflammatory Bowel Disease | Every 3 months up to 6 months, then every 6 months up to 24 months
  Baseline will be assessed as follows: Never Present, Positive History (Not present- Complete Remission,Time since remission onset; Present- Assessment of severity using a five point Likert scale (0 = Absent (Clear for Psoriasis); 5 = Most Severe)) Follow-up visits will be assessed as follows:Not present (Never present, Complete remission) Present (New Onset or Recurrence, Assessment of severity using a five point Likert scale (0 = Absent; 5 = Most Severe))
Occurrence, flare-up or exacerbation of Extra Articular Manifestations in Enthesitis of the Heel: Achilles Tendon and Plantar Fascia | Every 3 months up to 6 months, then every 6 months up to 24 months
  Baseline will be assessed as follows: Never Present, Positive History (Not present- Complete Remission,Time since remission onset; Present- Assessment of severity using a five point Likert scale (0 = Absent (Clear for Psoriasis); 5 = Most Severe)) Follow-up visits will be assessed as follows:Not present (Never present, Complete remission) Present (New Onset or Recurrence, Assessment of severity using a five point Likert scale (0 = Absent; 5 = Most Severe))

SECONDARY OUTCOMES:
BASFI (Bath AS Functional Assay) | Every 3 months up to 6 months, then every 6 months up to 24 months
  This is a 100 VAS with 0 indicating lowest functional limitations and 10 highest functional limitations
PASQ (Psoriasis and Arthritis Screening Questionnaire) | Every 3 months up to 6 months, then every 6 months up to 24 months
  This is an 11 item tool that ascertains self reported presence of joint pain and swelling.
BASDAI (Bath AS Disease Activity Index) | Every 3 months up to 6 months, then every 6 months up to 24 months
  This is a 100 VAS with 0 indicating lowest disease activity and 10 highest disease activity

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (56):
- Canada (56):
  - Rheumatology Clinic /ID# 54768, Calgary, Alberta
  - Associate Clinic /ID# 64274, Calgary, Alberta
  - Pont, Cranbrook, BC, CA /ID# 55242, Cranbrook, British Columbia
  - Dr. Barbara T. Blumenauer Inc. /ID# 55226, Kamloops, British Columbia
  - Hudson, Kamloops, Canada /ID# 54577, Kamloops, British Columbia
  - Dr. Maqbool R. Sheriff Inc. /ID# 55247, Nanaimo, British Columbia
  - Stewart, Penticton, CA /ID# 67096, Penticton, British Columbia
  - Dr. Michael Buchanan, Inc. /ID# 55227, Prince George, British Columbia
  - Dr. J. Antonio Avina-Zubieta /ID# 68263, Richmond, British Columbia
  - Dr. Alfonso Verdejo Inc. /ID# 54572, Vancouver, British Columbia
  - Dr. Milton F. Baker Inc. /ID# 55197, Victoria, British Columbia
  - Manitoba Clinic /ID# 54580, Winnipeg, Manitoba
  - Bulleid Henderson Prof. Corp. /ID# 55256, Fredericton, New Brunswick
  - Ecker, Fredericton, CA /ID# 54748, Fredericton, New Brunswick
  - Nexus Clinical Research /ID# 54757, St. John's, Newfoundland and Labrador
  - St. Clare's Mercy Hospital /ID# 54767, St. John's, Newfoundland and Labrador
  - Qe Ii Hsc /Id# 55261, Halifax, Nova Scotia
  - Dr. Juris Lazovskis Inc. /ID# 61562, Sydney, Nova Scotia
  - Pavlova, Hamilton, CA /ID# 65011, Ancaster, Ontario
  - Waterside Clinique /ID# 72174, Barrie, Ontario
  - Joshi, Brampton, Canada /ID# 54758, Brampton, Ontario
  - Brockville Medical Center /ID# 65502, Brockville, Ontario
  - Dr. Sanjay Dixit Medicine Professional Corporation /ID# 67347, Burlington, Ontario
  - Aviva Clinical Trial Group /ID# 54764, Burlington, Ontario
  - Dr. Chrisotomor Kouroukis & Dr /ID# 137831, Dundas, Ontario
  - Charlton Medical Centre /ID# 133072, Hamilton, Ontario
  - Charlton Medical Centre /ID# 55417, Hamilton, Ontario
  - Dr. William G. Bensen Centre /ID# 54762, Hamilton, Ontario
  - West Mountain Medical Center /ID# 128877, Hamilton, Ontario
  - KW Musculoskeletal Research /ID# 70093, Kitchener, Ontario
  - Brandusa Florica Med Prof Corp /ID# 81877, Mississauga, Ontario
  - Montgomery, Mississauga, CA /ID# 54581, Mississauga, Ontario
  - Credit Valley Rheumatology /ID# 54750, Mississauga, Ontario
  - Imtiaz MS Khan Medicine Prof /ID# 55401, Mississauga, Ontario
  - Morassut, Nepean, Canada /ID# 55410, Nepean, Ontario
  - The Arthritis Program Res Grp /ID# 54755, Newmarket, Ontario
  - Rajwinder S. Dhillon Medicine /ID# 138671, Niagara Falls, Ontario
  - Kapur, Ottawa, Canada /ID# 55397, Ottawa, Ontario
  - Davis, Ottawa, CA /ID# 55296, Ottawa, Ontario
  - Setty, Owen Sound, CA /ID# 54583, Owen Sound, Ontario
  - Niagara Peninsula Arthritis Ct /ID# 67282, St. Catharines, Ontario
  - Pedvis Med Prof Corp /ID# 55411, Toronto, Ontario
  - Hamilton, Toronto, CA /ID# 54575, Toronto, Ontario
  - Jonathan Stein Med Prof Corp /ID# 55451, Toronto, Ontario
  - Karasik, Toronto, CA /ID# 54751, Toronto, Ontario
  - Dr. Samuel K Silverberg /ID# 55449, Toronto, Ontario
  - Ctr de Med Sportive de Laval /ID# 54576, Laval, Quebec
  - Institut de Rhum. de Montreal /ID# 54761, Montreal, Quebec
  - Jewish General Hospital /ID# 63655, Montreal, Quebec
  - PSS Medical Inc. /ID# 54754, Montreal, Quebec
  - Couture, Outremont, CA /ID# 54574, Outremont, Quebec
  - Ctr. de Rheum de l'est du QC /ID# 54765, Rimouski, Quebec
  - Clinique Medicale Langelier /ID# 55460, Saint-Léonard, Quebec
  - Groupe de Recherche en Maladies Osseuses /ID# 45623, Sainte-Foy, Quebec
  - Ctr. de Recherche Musculo-Sque /ID# 55469, Trois-Rivières, Quebec
  - Rheum Disease Ctr of Montreal /ID# 143963, Westmount, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P12-672.pdf